CLINICAL TRIAL: NCT00005185
Title: Myocardial Infarction and Non-contraceptive Estrogen Use
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1063; R01HL032174 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Menopause; Postmenopause
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction

SUMMARY:
To evaluate whether the use of noncontraceptive estrogen influenced the incidence of first myocardial infarction in women.

DETAILED DESCRIPTION:
BACKGROUND:

The use of noncontraceptive estrogens declined after evidence was published that they increase the risk of endometrial cancer. Nonetheless, they are still used commonly and for long periods, especially by hysterectomized women. Use of the drugs has increased recently, perhaps because the drugs have been recommended as prophylaxis against osteoporosis. The drugs are also being promoted for use in conjunction with a progestin, because it is thought that the combination may protect against endometrial cancer. Little is known about the effects of these drug regimens on myocardial infarction risk, and some progestins (in particular the 19-norprogestins) are thought to influence lipid profiles unfavorably. Insofar as myocardial infarction is a major cause of morbidity and mortality in women beyond age 49, an effect of these drugs, either beneficial or adverse, on myocardial infarction risk is of considerable public health importance.

DESIGN NARRATIVE:

The design was that of a case-control study. Cases were selected from women admitted for the first episode of myocardial infarction to any of the participating hospitals in the Boston area. For each case, a control was selected from town lists of women living in the same neighborhood as the case and in the same five year age group. Cases were interviewed by telephone after discharge from the hospital, and the corresponding control was interviewed within a week or two of the case interview.

Information was obtained on: the timing and duration of non-contraceptive estrogen use, the names of the preparations and reasons for starting and stopping each episode of use; other drug use particularly oral contraceptives, aspirin, phenylpropanolamine; age at menopause; cigarette smoking; height and weight; histories of previous myocardial infarction, hypertension, pre-eclamptic toxemia, diabetes mellitus, angina pectoris and abnormal serum lipids; reproductive history; alcohol and coffee consumption; personality type based on the Framingham Type A Scale; family history of myocardial infarction; exercise; socioeconomic and life style factors; number of physician visits in last two years and total number of hospital admissions.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1986-04; Study Completion 1990-03 (Actual)

REFERENCES:
- [Background] Palmer JR, Rosenberg L, Shapiro S. "Low yield" cigarettes and the risk of nonfatal myocardial infarction in women. N Engl J Med. 1989 Jun 15;320(24):1569-73. doi: 10.1056/NEJM198906153202401. PMID 2725598
- [Background] Rosenberg L, Palmer JR, Shapiro S. Decline in the risk of myocardial infarction among women who stop smoking. N Engl J Med. 1990 Jan 25;322(4):213-7. doi: 10.1056/NEJM199001253220401. PMID 2294448
- [Background] Rosenberg L, Palmer JR, Lesko SM, Shapiro S. Oral contraceptive use and the risk of myocardial infarction. Am J Epidemiol. 1990 Jun;131(6):1009-16. doi: 10.1093/oxfordjournals.aje.a115592. PMID 2343853
- [Background] Palmer JR, Rosenberg L, Shapiro S. Stature and the risk of myocardial infarction in women. Am J Epidemiol. 1990 Jul;132(1):27-32. doi: 10.1093/oxfordjournals.aje.a115639. PMID 2356811
- [Background] Palmer JR, Rosenberg L, Shapiro S. Reproductive factors and risk of myocardial infarction. Am J Epidemiol. 1992 Aug 15;136(4):408-16. doi: 10.1093/oxfordjournals.aje.a116513. PMID 1415160
- [Background] Palmer JR, Rosenberg L, Rao RS, Shapiro S. Coffee consumption and myocardial infarction in women. Am J Epidemiol. 1995 Apr 15;141(8):724-31. doi: 10.1093/oxfordjournals.aje.a117494. PMID 7709915
- [Background] Rosenberg L, Palmer JR, Shapiro S. A case-control study of myocardial infarction in relation to use of estrogen supplements. Am J Epidemiol. 1993 Jan 1;137(1):54-63. doi: 10.1093/oxfordjournals.aje.a116602. PMID 8434573